CLINICAL TRIAL: NCT00531635
Title: Induction of Mixed Hemopoietic Chimerism in Patients Using Fludarabine, Low Dose TBI, PBSC Infusion and Post Transplant in Immunosuppression w/CSA & Mycophenolate Mofetil
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC#2001-051
Record Dates: First submitted 2007-09-17; First posted 2007-09-19 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Post Transplant in Immunosuppression w/CSA & Mycophenolate Mofetil
Keywords: Mixed hemopoietic chimerism, Fludarabine, TBI, PBSC, immunosuppression, Mycophenolate Mofetil
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Induction of Mixed Hemopoietic Chimerism in Patients Using Mycophenolate Mofetil

SUMMARY:
Induction of mixed hemopoietic chimerism in patients using Fludarabine, Low Dose TBI, PBSC Infusion and post transplant in immunosuppression w/CSA & Mycophenolate Mofetil

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving Fludarabine, Low Dose TBI, PBSC Infusion and post transplant in immunosuppression w/CSA & Mycophenolate Mofetil.

Exclusion Criteria:

* Uncontrolled major medical illnesses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2002-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 2001-2012

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Aljurf, MD, Principal Investigator — KFSH&RC
Locations (1):
- KFSH&RC, Riyadh, Saudi Arabia